CLINICAL TRIAL: NCT04020692
Title: Home Improvement Initiative of the TRaitement Optimisé Medicamenteux After Hospitalization
Acronym: IATRO'MED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Delays were caused by the covid-19 pandemic and a lack of staff on the saint vincent hospital site to take charge of the study
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 7363
Record Dates: First submitted 2019-07-09; First posted 2019-07-16 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Older Adult; Chronic Disease; Clinical Pharmacy; Surgery; Ambulatory Care
Keywords: Multicenter study; Before-and-after type study; Minimal risks and constraints
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Intervention Model Description: The issue of drug continuity after hospital discharge has become a major issue in recent years. When patients return home, the drugs taken do not correspond to the treatments prescribed at the end of the hospitalization. This is due to appropriate or inappropriate initiatives of the patients (or their relatives) and/or the physicians accompanying them. Prescribed medications, on the other hand, are almost always dispensed by community pharmacists.
  The scope chosen in this project is that the intervention of an operational clinical pharmacy team (EOPC), targeting both patient and health care professionals (inpatient and outpatient), will maintain, in outpatient care, the drugs treatments that have been optimized during hospitalization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- "intervention " group (Experimental): Patient At D0, the patient receives his discharge drugs prescription and benefits from a pharmaceutical counselling.
  At D+3, he benefits from a telephone follow-up (good understanding of the methods of taking drugs, collection of difficulties).
  Community pharmacist At D0, he receives the discharge drugs prescription. At D+3, he is contacted to collect information relating to drugs 'dispensation.
  The attending physician At D0, he is informed of the patient's discharge and his drugs treatment
  At D45, the data collection is based on telephone interviews [attending physician, pharmacist and patient (and if applicable the caregiver)].
  It makes possible to collect drugs taken by the patient as well as significant events over the period (acute pathologies, re-hospitalizations, etc.).
  Interventions: Behavioral: EOPC Intervention
- Control group (No Intervention): At D0, the patient receives his discharge drugs prescription.
  At D45, the data collection is based on telephone interviews [attending physician, pharmacist and patient (and if applicable the caregiver)].
  It makes possible to collect drugs taken by the patient as well as significant events over the period (acute pathologies, re-hospitalizations, etc.).

INTERVENTIONS:
Behavioral: EOPC Intervention — The issue of drug continuity after hospital discharge has become a major issue in recent years. When patients return home, the drugs taken do not correspond to the treatments prescribed at the end of the hospitalization. This is due to appropriate or inappropriate initiatives of the patients (or their relatives) and/or the physicians accompanying them. Prescribed medications, on the other hand, are almost always dispensed by community pharmacists.
  The scope chosen in this project is that the intervention of an operational clinical pharmacy team (EOPC), targeting both patient and health care professionals (inpatient and outpatient), will maintain, in outpatient care, the drugs treatments that have been optimized during hospitalization.
  Arms: "intervention " group

SUMMARY:
The hypothesis is that the intervention of an operational clinical pharmacy team (EOPC), targeting both patients and hospital and health care professionals, allows: i) to initiate a therapeutic review during hospitalization, ii) to accompany the patients upon hospital discharge, iii) to maintain, in outpatient care, the drug treatments that have been optimized during hospitalization.

The main objective of the study is to demonstrate that the intervention of an EOPC in surgical departments and then in outpatient care makes it possible to maintain, 45 days after the discharge of the patients aged 65 years and over, the chronic outpatient treatments revised and optimized during the hospital stay.

The secondary objectives are to measure the impacts of EOPC's intervention on:

* unexpected readmissions, emergency use, medical complications and adverse drug reactions;
* patient and health professional satisfactions (community pharmacists and physicians);
* the costs of drug treatments in ambulatory care.

ELIGIBILITY:
Inclusion Criteria:

* Patient (man or woman)
* age ≥ 65 years with more than 3 drugs taken for 3 months, stay in surgery with a duration of ≥ 1 days including urgent surgery;
* affiliated to a social health insurance scheme;
* for whom a return home is possible;
* able to understand the objectives of the research and give informed, dated and signed consent.

Exclusion Criteria:

* Patient (man or woman)
* with as a hospital discharge an entry into a nursing home or long-term care called "important medical and technical care (SMTI);
* with cognitive or other problems preventing consent (at the discretion of the geriatric expertise team);
* under the safeguard of justice;
* under tutorship or curatorship.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 223 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-02-02 (Actual)

PRIMARY OUTCOMES:
Compliance of patients' medication intake at 45 days (D45) compared to the discharge prescription (D0): drugs prescribed and taken by patients (chronic disease treatments only) | 45 days
  Compliance is defined as the absence of discrepancies between D0 and D+45. Conversely, the presence of a discrepancy is defined as the presence of at least one deviation of drug intake at D+45 from D0.

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Groupe Hospitalier Saint Vincent, Strasbourg
  - Les Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: Undecided